CLINICAL TRIAL: NCT06358053
Title: A Phase I Study to Evaluate the Safety, Tolerance and Efficacy of CRTE7A2-01 TCR-T Cells in HLA-A*02:01+ Subjects With HPV16 Positive Advanced Cervical, Anal, or Head and Neck Cancers and Other Solid Tumors
Brief Title: CRTE7A2-01 TCR-T Cells for HPV-16 Positive Advanced Cancers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Corregene Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRTE7A2-2302C
Record Dates: First submitted 2024-04-02; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Cervical Cancer; Anal Cancer; Head and Neck Cancers; Other Solid Tumors
Keywords: HPV; E7; immunotherapy; T cell; Adoptive cell therapy; T cell receptor; TCR
MeSH Terms: conditions — Uterine Cervical Neoplasms; Anus Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CRTE7A2-01 TCR-T cell therapy (Experimental): This study is a single-arm Phase I study, encompassing both dose escalation and dose expansion phases. Patients will undergo lymphocytapheresis, then treatment with TCR-T cell (at escalating doses) + IL-2
  Interventions: Drug: CRTE7A2-01 TCR-T cell therapy

INTERVENTIONS:
Drug: CRTE7A2-01 TCR-T cell therapy — Drug 1: Fludarabine + Cyclophosphamide Drug 2: Interleukin-2 Drug 3: CRTE7A2-01 TCR-T Cell
  Other Names: CRTE7A2

SUMMARY:
A single center, open, single arm dose escalation and dose expansion phase I study to evaluate the safety, tolerability, and efficacy of CRTE7A2-01 TCR-T cells in HLA-A*02:01+ Subjects HPV16 positive advanced cervical, anal, or head and neck cancers. The study will determine RP2D of CRTE7A2-01 TCR-T cell injection.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years and 65 years. 2. Patients with advanced solid tumors (such as cervical cancer, head and neck tumors, anal cancer, and other malignancies) who have failed standard treatment confirmed by histology and/or cytology, or who are intolerant to such treatment, and for whom there is no effective therapy available after standard treatment failure are considered as end-stage patients. Specifically for:

1. Cervical cancer: a) Patients who have previously failed at least second-line systemic therapy (including at least one platinum-based regimen or anti-angiogenic therapy) and have shown disease progression or intolerance confirmed by pathological or radiological examination during or after the most recent treatment course, and are not amenable to treatment with surgery or radiotherapy, with no standard treatment options currently available for recurrent or metastatic cervical cancer.
2. Nasopharyngeal cancer: a) Patients who have previously failed at least third-line systemic therapy or are intolerant, not amenable to treatment with surgery or radiotherapy, with no standard treatment options currently available for recurrent or metastatic nasopharyngeal cancer; b) EB virus negative.
3. Head and neck squamous cell carcinoma: a) Patients who have previously failed at least second-line systemic therapy or are intolerant, with no standard treatment options currently available for recurrent or metastatic head and neck squamous cell carcinoma (non-nasal).

3. Confirmation of HPV16 positive and HLA-A*02:01 allele. 4. ECOG performance status of 0-1. 5. Estimated life expectancy ≥ 3 months. 6. Patients must have at least one measurable lesion defined by RECIST 1.1. 7. Female patients of childbearing age must undergo a serum pregnancy test within 7 days prior to study treatment and the results must be negative, and are willing to use a very effective and reliable method of contraception from screening through 6 months after the last dose of study treatment.

8. The patient must be willing to sign the informed consent form and have a good anticipation of compliance with study procedure.

Exclusion Criteria:

1. Patient received any genetically modified T cell therapy.
2. Patient is being treated with T cell immunosuppressive agent （such as cyclophosphamide, FK506,tripterygium glycosides） or T cell immunoagonist.
3. Patients received chemotherapy, targeted therapy, immunotherapy, or other investigational agents within 2 weeks and received radiotherapy within 4 weeks before apheresis.
4. Patients have any organ system function impairment as defined below:

   * leukocytes<3.0 x 109/L
   * absolute neutrophil count >1.5 x 109/L
   * hemoglobin<90g/L
   * platelets <100 x 1010/L
   * lymphocytes<0.5 x 109/L
   * percentage of lymphocytes<15%
   * creatinine>1.5×ULN or creatinine clearance <50mL/min
   * total bilirubin>3×ULN; ALT/AST>3×ULN (patients with liver metastasis,>5×ULN)
   * INR>1.5×ULN; APTT>1.5×ULN
   * SpO2≤90%

6. Patinets has serious medical conditions, disorders, and / or comorbidities, including, but are not limited to: severe heart disease, cerebrovascular disease, epileptic seizures, uncontrolled diabetes (CTCAE 5.0: FBG ≥ 2 grade), active infection, active digestive tract Ulcer, gastrointestinal bleeding, intestinal obstruction, pulmonary fibrosis, renal failure, respiratory failure.

7. Patient has a severe cardiovascular disease with 6 months before screening, including, but are not limited to, myocardial infarction, severe or unstable angina, coronary or peripheral artery bypass grafting, Heart failure NYHA grade Ⅲ or Ⅳ.

8. Left Ventricular Ejection Fractions (LVEF) <50%. 9. Patient has a known active brain metastases. 10. Patient has a known myelodysplastic syndrome (MDS) or lymphoma. 11. Patient has a known active autoimmune disease, including , but are not limited to, acquired or congenital immunodeficiency disease, allogeneic organ transplantation, autoimmune hepatitis, systemic lupus erythematosus, inflammatory bowel disease.

12. Patient has a known active Hepatitis B or Hepatitis C. 13. Patient has a history of Human Immunodeficiency Virus (HIV) . 14. Patient has a history of syphilis. 15. Pregnant or lactating women. 16. Patient has a known active mental and neurological diseases. 17. The principal investigator judged that it is not suitable to participate in this clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
DLT | 28 days
  Dose-limiting toxicity
RP2D | 2 years
  Recommended Phase 2 Dose
cevents (SAEs). | 2 years
  Incidence of treatment related AEs, AEs of special interest and serious adverse events (SAEs).

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 2 years
  Assessed by RECIST 1.1
Disease Control Rate (DCR) | 2 years
  Assessed by RECIST 1.1
Duration of Response (DOR) | 2 years
  Assessed by RECIST 1.1
Progression-Free Survival (PFS) | 2 years
  Assessed by RECIST 1.1
Overall Survival(OS) | 2 years
  Assessed by RECIST 1.1

OTHER OUTCOMES:
Peripheral blood TCR-T cell copy number | 2 years
  Peripheral blood TCR-T cell copy number

CONTACTS AND LOCATIONS:
Overall Officials: Yang Xiang, Doctor, Principal Investigator — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: No